CLINICAL TRIAL: NCT00735280
Title: Non-randomized, Open-label, Historical Control, Single Group Assignment Trial of a Reduced Dose of Unfractionated Heparin in Patients Undergoing Percutaneous Coronary Interventions
Brief Title: Reduced Dose of Unfractionated Heparin in Patients Undergoing PCI
Acronym: ISAR-REACT-3A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. A01408
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease, stent, heparin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced dose of unfractionated heparin (Experimental)
  Interventions: Drug: unfractionated heparin

INTERVENTIONS:
Drug: unfractionated heparin — bolus of 100 U/kg of unfractionated heparin

SUMMARY:
The aim of this trial is to evaluate whether a reduction in the heparin dose from 140 to 100 U/kg is associated with a better net clinical outcome in patients undergoing PCI after pretreatment with 600mg clopidogrel

DETAILED DESCRIPTION:
Percutaneous coronary interventions, mostly with implantation of bare-metal or drug-eluting stents, are commonly used to treat patients with coronary artery disease. Various periprocedural adjunct antithrombotic therapies have been investigated and are being used. Unfractionated heparin (UFH) has been the standard adjunctive antithrombin therapy during PCI for more than 25 years. Combined antiplatelet treatment consisting of aspirin and a thienopyridine has significantly reduced early ischaemic events following coronary stenting (1). Thienopyridines act by irreversibly inhibiting the platelet adenosine diphosphate (ADP) P2Y12 receptor. Compared to ticlopidine, clopidogrel has the advantage of a more favourable side effect profile (2) and more rapid onset of action.(3,4) Pretreatment with a loading dose of 300mg clopidogrel improved outcomes (5-7) and is recommended by current guidelines for patients undergoing PCI. (8) More recently, trials have shown that the larger loading dose of 600mg achieves more rapid and more potent inhibition of platelet aggregation than 300 mg do.(9-11) The results of several randomized controlled trials suggest that pretreatment with 600mg clopidogrel might obviate the need for IIb/IIIa inhibitors in a broad spectrum of patients undergoing PCI (12-14) although no formal direct comparison of different clopidogrel doses has been assessed by trials sufficiently powered for clinical endpoints. The Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment (ISAR-REACT) trial showed that after pretreatment with 600mg clopidogrel for at least 2 hours before the intervention, additional use of abciximab was not associated with any clinically measurable benefit among low-to-intermediate risk patients who underwent PCI.(12) Even in higher risk settings such as small vessel size (14) and the presence of diabetes (13)additional use of abciximab was not associated with a measurable clinical benefit in patients pretreated with 600mg clopidogrel. An important exception is the group of patients with non-ST-segment elevation ACS. In the ISAR-REACT-2 trial that enrolled this category of patients those with an elevated troponin level did benefit from abciximab even after pretreatment with 600mg clopidogrel.(15) The recently completed ISAR-REACT-3 trial compared unfractionated heparin with the direct thrombin inhibitor bivalirudin in biomarker negative patients with stable and unstable angina undergoing contemporary PCI. Bivalirudin did not provide "net clinical benefit" - did not reduce the quadruple endpoint - at 30 days compared to unfractionated heparin. However, there was a significant reduction in bleeding with bivalirudin (16) The heparin dose regimen used in ISAR-REACT-3 diverges from current US practice insofar as the majority of patients received a bolus dose of 140 U/kg with no follow up ACT measurement and no additional heparin doses. Although heparin has been the standard antithrombin therapy in interventional cardiology for decades, its optimal dose is still not known. During the last years there has been a trend towards using lower heparin doses. In most interventional trials in the United States it is now current practice to use a bolus of not more than 100 U/kg. (8) Many interventionalists believe that a dose lower than 140 U/kg is associated with a better clinical outcome. However, no studies have been performed to identify the most appropriate dose of heparin. Since pretreatment with clopidogrel has proven to reduce ischemic events, a heparin dose of 140U/kg might conceivably be too high. A lower dose might prove to be as effective in preventing ischemic endpoints while reducing the risk of bleeding if patients were pretreated with 600mg clopidogrel prior to the intervention. Therefore the aim of this trial is to evaluate whether a reduction in the heparin dose from 140 to 100 U/kg is associated with a better net clinical outcome in patients undergoing PCI after pretreatment with 600mg clopidogrel. The hypothesis to be tested is whether a reduced dose of 100U/kg heparin is superior to the higher dose of 140U/kg used in the ISAR-REACT-3 trial (historical control) regarding the combined incidence of death, myocardial infarction, urgent target vessel revascularization within 30 days and in hospital major bleeding. The ISAR-REACT-3a trial will enroll a patient population with a similar risk profile to that of patients included in ISAR-REACT-3. Biomarker negative patients with stable or unstable angina undergoing PCI will receive a reduced dose heparin bolus of 100U/kg. Results will be compared with the ISAR-REACT-3 trial (historical control). Primary comparison will be with the heparin arm of ISAR-REACT-3 regarding the primary endpoint ("Net clinical benefit", the combined incidence of death, myocardial infarction, urgent target vessel revascularization within 30 days and in hospital major bleeding). A secondary aspect will be the comparison with the historical bivalirudin group of the ISAR-REACT-3 trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years undergoing a PCI procedure
2. Pretreatment with 600mg clopidogrel at least 2 hours before the intervention
3. Informed, written consent by the patient or her/his legally-authorized representative for participation in the study.

Exclusion Criteria:

1. Recent ST-elevation myocardial infarction within the last 48 hours
2. Acute coronary syndromes with positive biomarkers (Troponin T > 0.03 μg/L or CK-MB > ULN)
3. Cardiogenic shock
4. Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than one year or that may result in protocol non-compliance
5. Active bleeding; bleeding diathesis
6. History of gastrointestinal or genitourinary bleeding within the last 6 weeks
7. Presence of diseases which have a high probability of vascular lesions and subsequent bleeding such as active gastric ulcer or active ulcerous colitis
8. Recent trauma or major surgery in the last month
9. Ophthalmic surgery or brain surgery in the last month
10. Retinopathies or vitreous body bleeding in the last month
11. History of intracranial bleeding or structural abnormalities (for example aneurysm of cerebral arteries)
12. Suspected aortic dissection; pericarditis and subacute bacterial endocarditis
13. Patient's refusal to blood transfusion.
14. Oral anticoagulation therapy with coumarin derivative within the last 7 days
15. Treatment with UFH within 6 hours unless an ACT is less than 150 sec or low-molecular weight heparin within 8 hours before enrollment
16. Treatment with bivalirudin within 24 hours before enrollment
17. Severe uncontrolled hypertension >180/110 mmHg unresponsive to therapy
18. Planned staged PCI procedure within 30 days from index procedure or prior PCI within the last 30 days.
19. Relevant hematologic deviations: hemoglobin < 100 g/L, platelet count < 100 x 109 /L.
20. Glomerular filtration rate (GFR) < 30 ml/min or serum creatinine > 30 mg/L or dependence on renal dialysis.
21. Known allergy to the study medications: aspirin, clopidogrel, UFH, true anaphylaxis after prior exposure to contrast media.
22. Known heparin-induced thrombocytopenia (Typ II)
23. Previous enrollment in this trial.
24. Pregnancy (present, suspected or planned) or positive pregnancy test.
25. Spinal, peridural and epidural anesthesia
26. Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2505 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be a composite of death, MI, urgent TVR after 30 days or in hospital bleeding (quadruple endpoint, "net clinical benefit"). | 30 days

SECONDARY OUTCOMES:
Composite of death, MI or urgent TVR (Triple endpoint to assess ischemic complications) | 30 days
Composite of death, MI or TVR | 1 year after the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum München; Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (3):
- Germany (3):
  - Herz-Zentrum, Bad Krozingen
  - Deutsches Herzzentrum München, München
  - Klinikum rechts der Isar der Technischen Universität München, München

REFERENCES:
- [Background] Schomig A, Neumann FJ, Kastrati A, Schuhlen H, Blasini R, Hadamitzky M, Walter H, Zitzmann-Roth EM, Richardt G, Alt E, Schmitt C, Ulm K. A randomized comparison of antiplatelet and anticoagulant therapy after the placement of coronary-artery stents. N Engl J Med. 1996 Apr 25;334(17):1084-9. doi: 10.1056/NEJM199604253341702. PMID 8598866
- [Background] Bertrand ME, Rupprecht HJ, Urban P, Gershlick AH; CLASSICS Investigators. Double-blind study of the safety of clopidogrel with and without a loading dose in combination with aspirin compared with ticlopidine in combination with aspirin after coronary stenting : the clopidogrel aspirin stent international cooperative study (CLASSICS). Circulation. 2000 Aug 8;102(6):624-9. doi: 10.1161/01.cir.102.6.624. PMID 10931801
- [Background] Thebault JJ, Kieffer G, Cariou R. Single-dose pharmacodynamics of clopidogrel. Semin Thromb Hemost. 1999;25 Suppl 2:3-8. PMID 10440415
- [Background] Gawaz M, Seyfarth M, Muller I, Rudiger S, Pogatsa-Murray G, Wolf B, Schomig A. Comparison of effects of clopidogrel versus ticlopidine on platelet function in patients undergoing coronary stent placement. Am J Cardiol. 2001 Feb 1;87(3):332-6, A9. doi: 10.1016/s0002-9149(00)01369-2. PMID 11165971
- [Background] Steinhubl SR, Berger PB, Mann JT 3rd, Fry ET, DeLago A, Wilmer C, Topol EJ; CREDO Investigators. Clopidogrel for the Reduction of Events During Observation. Early and sustained dual oral antiplatelet therapy following percutaneous coronary intervention: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2411-20. doi: 10.1001/jama.288.19.2411. PMID 12435254
- [Background] Chan AW, Moliterno DJ, Berger PB, Stone GW, DiBattiste PM, Yakubov SL, Sapp SK, Wolski K, Bhatt DL, Topol EJ; TARGET Investigators. Triple antiplatelet therapy during percutaneous coronary intervention is associated with improved outcomes including one-year survival: results from the Do Tirofiban and ReoProGive Similar Efficacy Outcome Trial (TARGET). J Am Coll Cardiol. 2003 Oct 1;42(7):1188-95. doi: 10.1016/s0735-1097(03)00944-6. PMID 14522478
- [Background] Assali AR, Salloum J, Sdringola S, Moustapha A, Ghani M, Hale S, Schroth G, Fujise K, Anderson HV, Smalling RW, Rosales OR. Effects of clopidogrel pretreatment before percutaneous coronary intervention in patients treated with glycoprotein IIb/IIIa inhibitors (abciximab or tirofiban). Am J Cardiol. 2001 Oct 15;88(8):884-6, A6. doi: 10.1016/s0002-9149(01)01897-5. No abstract available. PMID 11676953
- [Background] Smith SC Jr, Feldman TE, Hirshfeld JW Jr, Jacobs AK, Kern MJ, King SB 3rd, Morrison DA, O'Neil WW, Schaff HV, Whitlow PL, Williams DO, Antman EM, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; ACC/AHA/SCAI Writing Committee to Update 2001 Guidelines for Percutaneous Coronary Intervention. ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/SCAI Writing Committee to Update 2001 Guidelines for Percutaneous Coronary Intervention). Circulation. 2006 Feb 21;113(7):e166-286. doi: 10.1161/CIRCULATIONAHA.106.173220. No abstract available. PMID 16490830
- [Background] Montalescot G, Sideris G, Meuleman C, Bal-dit-Sollier C, Lellouche N, Steg PG, Slama M, Milleron O, Collet JP, Henry P, Beygui F, Drouet L; ALBION Trial Investigators. A randomized comparison of high clopidogrel loading doses in patients with non-ST-segment elevation acute coronary syndromes: the ALBION (Assessment of the Best Loading Dose of Clopidogrel to Blunt Platelet Activation, Inflammation and Ongoing Necrosis) trial. J Am Coll Cardiol. 2006 Sep 5;48(5):931-8. doi: 10.1016/j.jacc.2006.04.090. Epub 2006 Aug 17. PMID 16949482
- [Background] Price MJ, Coleman JL, Steinhubl SR, Wong GB, Cannon CP, Teirstein PS. Onset and offset of platelet inhibition after high-dose clopidogrel loading and standard daily therapy measured by a point-of-care assay in healthy volunteers. Am J Cardiol. 2006 Sep 1;98(5):681-4. doi: 10.1016/j.amjcard.2006.03.054. Epub 2006 Jul 7. PMID 16923461
- [Background] von Beckerath N, Taubert D, Pogatsa-Murray G, Schomig E, Kastrati A, Schomig A. Absorption, metabolization, and antiplatelet effects of 300-, 600-, and 900-mg loading doses of clopidogrel: results of the ISAR-CHOICE (Intracoronary Stenting and Antithrombotic Regimen: Choose Between 3 High Oral Doses for Immediate Clopidogrel Effect) Trial. Circulation. 2005 Nov 8;112(19):2946-50. doi: 10.1161/CIRCULATIONAHA.105.559088. Epub 2005 Oct 31. PMID 16260639
- [Background] Kastrati A, Mehilli J, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Bollwein H, Volmer C, Gawaz M, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. A clinical trial of abciximab in elective percutaneous coronary intervention after pretreatment with clopidogrel. N Engl J Med. 2004 Jan 15;350(3):232-8. doi: 10.1056/NEJMoa031859. PMID 14724302
- [Background] Mehilli J, Kastrati A, Schuhlen H, Dibra A, Dotzer F, von Beckerath N, Bollwein H, Pache J, Dirschinger J, Berger PP, Schomig A; Intracoronary Stenting and Antithrombotic Regimen: Is Abciximab a Superior Way to Eliminate Elevated Thrombotic Risk in Diabetics (ISAR-SWEET) Study Investigators. Randomized clinical trial of abciximab in diabetic patients undergoing elective percutaneous coronary interventions after treatment with a high loading dose of clopidogrel. Circulation. 2004 Dec 14;110(24):3627-35. doi: 10.1161/01.CIR.0000148956.93631.4D. Epub 2004 Nov 7. PMID 15531766
- [Background] Hausleiter J, Kastrati A, Mehilli J, Schuhlen H, Pache J, Dotzer F, Glatthor C, Siebert S, Dirschinger J, Schomig A; ISAR-SMART-2 Investigators. A randomized trial comparing phosphorylcholine-coated stenting with balloon angioplasty as well as abciximab with placebo for restenosis reduction in small coronary arteries. J Intern Med. 2004 Nov;256(5):388-97. doi: 10.1111/j.1365-2796.2004.01398.x. PMID 15485474
- [Background] Kastrati A, Mehilli J, Neumann FJ, Dotzer F, ten Berg J, Bollwein H, Graf I, Ibrahim M, Pache J, Seyfarth M, Schuhlen H, Dirschinger J, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic: Regimen Rapid Early Action for Coronary Treatment 2 (ISAR-REACT 2) Trial Investigators. Abciximab in patients with acute coronary syndromes undergoing percutaneous coronary intervention after clopidogrel pretreatment: the ISAR-REACT 2 randomized trial. JAMA. 2006 Apr 5;295(13):1531-8. doi: 10.1001/jama.295.13.joc60034. Epub 2006 Mar 13. PMID 16533938
- [Background] Kastrati A, Neumann FJ, Mehilli J, Byrne RA, Iijima R, Buttner HJ, Khattab AA, Schulz S, Blankenship JC, Pache J, Minners J, Seyfarth M, Graf I, Skelding KA, Dirschinger J, Richardt G, Berger PB, Schomig A; ISAR-REACT 3 Trial Investigators. Bivalirudin versus unfractionated heparin during percutaneous coronary intervention. N Engl J Med. 2008 Aug 14;359(7):688-96. doi: 10.1056/NEJMoa0802944. PMID 18703471
- [Derived] Schulz S, Mehilli J, Neumann FJ, Schuster T, Massberg S, Valina C, Seyfarth M, Pache J, Laugwitz KL, Buttner HJ, Ndrepepa G, Schomig A, Kastrati A; Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 3A Trial Investigators. ISAR-REACT 3A: a study of reduced dose of unfractionated heparin in biomarker negative patients undergoing percutaneous coronary intervention. Eur Heart J. 2010 Oct;31(20):2482-91. doi: 10.1093/eurheartj/ehq330. Epub 2010 Aug 30. PMID 20805113